CLINICAL TRIAL: NCT01526122
Title: A PhaseⅠ Study to Compare the Pharmacokinetic Characteristics and Safety After Oral Administration of G0041(75/100mg) With Those of Clopidogrel 75mg & Aspirin 100mg Coadministration in Healthy Male Volunteers
Brief Title: Pharmacokinetics & Safety Study of Clopidogrel 75mg and Aspirin 100mg Coadministration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: G0041(75/100mg)_AS_Ⅰ
Record Dates: First submitted 2012-01-11; First posted 2012-02-03 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Atherosclerosis
Keywords: Clopidogrel; Aspirin; coadministration
MeSH Terms: conditions — Atherosclerosis | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G0041(75/100mg) (Experimental)
  Interventions: Drug: G0041(75/100mg)
- Clopidogrel & Aspirin (Active Comparator)
  Interventions: Drug: Clopidogrel & Aspirin

INTERVENTIONS:
Drug: G0041(75/100mg) — G0041(75/100mg) 2 capsules(Clopidogrel 75mg & Aspirin 100mg in 1 capsule), PO
  Arms: G0041(75/100mg)
Drug: Clopidogrel & Aspirin — Clopidogrel 75mg 2 tablets & Aspirin 100mg 2 capsules, PO
  Arms: Clopidogrel & Aspirin

SUMMARY:
The purpose of this study is to compare characteristics and safety after oral administration of G0041(75/100mg) 2 tablets with those of Clopidogrel 75mg 2 tablets & Aspirin 100mg 2 capsules coadministration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy male volunteers between the ages of 20 to 50 years old
* weight more than 55kg and within the range of ±20% of IBW
* having neither congenital/chronic diseases nor pathological symptoms/findings as results of medical examination
* doctor determines to be suitable as subjects within 3 weeks ago before administration

Exclusion Criteria:

* Hypersensitivitiy(or history of hypersensitivity) to aspirin and clopidogrel
* Active Liver Diseases or exceed 1.5 times the normal range of AST, ALT, total bilirubin
* Exceed the normal range of PT, aPTT, BT & platelet counts under 150,000/㎣ or exceed 350,000/㎣
* Creatinine clearance < 80 mL/min
* Gastrointestinal diseases or surgeries that affect absorption of drug
* Congenital galactose intolerance, lactase deficiency and glucose-galactose malabsorption
* Excessive drinking(exceed 21units/week)
* Smoking over 10 cigarettes per day

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
C(max) of Clopidogrel | 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24h
AUC(last) of Clopidogrel | 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24h
C(max) of Acetylsalicylic acid | 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24h
AUC(last) of Acetylsalicylic acid | 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24h

SECONDARY OUTCOMES:
C(max) of Salicylic acid | 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24h
AUC(last) of Salicylic acid | 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 24h

CONTACTS AND LOCATIONS:
Overall Officials: Young-ran Yoon, M.D., Ph.D., Principal Investigator — Kyungpook National University Hospital

REFERENCES:
- [Background] Di Girolamo G, Czerniuk P, Bertuola R, Keller GA. Bioequivalence of two tablet formulations of clopidogrel in healthy Argentinian volunteers: a single-dose, randomized-sequence, open-label crossover study. Clin Ther. 2010 Jan;32(1):161-70. doi: 10.1016/j.clinthera.2010.01.010. PMID 20171421
- [Background] Bae SK, Seo KA, Jung EJ, Kim HS, Yeo CW, Shon JH, Park KM, Liu KH, Shin JG. Determination of acetylsalicylic acid and its major metabolite, salicylic acid, in human plasma using liquid chromatography-tandem mass spectrometry: application to pharmacokinetic study of Astrix in Korean healthy volunteers. Biomed Chromatogr. 2008 Jun;22(6):590-5. doi: 10.1002/bmc.973. PMID 18254152
- [Background] Kim SD, Kang W, Lee HW, Park DJ, Ahn JH, Kim MJ, Kim EY, Kim SW, Nam HS, Na HJ, Yoon YR. Bioequivalence and tolerability of two clopidogrel salt preparations, besylate and bisulfate: a randomized, open-label, crossover study in healthy Korean male subjects. Clin Ther. 2009 Apr;31(4):793-803. doi: 10.1016/j.clinthera.2009.04.017. PMID 19446152
- [Background] EMEA(2009), CHMP assessment report of DuoCover. EMEA/H/C/001144